CLINICAL TRIAL: NCT05429723
Title: A Randomized, Double-Blind, Placebo Controlled, Phase I Study to Assess, Safety, Tolerability, Pharmacokinetics of HS-10383 Administered Orally in China Healthy Adult Subjects
Brief Title: First-in-Human Study to Investigate the Safety and Tolerability and Pharmacokinetics of HS-10383
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10383-101
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cough
Keywords: RUCC, P2X3
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10383 (Experimental): HS-10383 was administered at 8 am on the first day, 4 dose levels
  Interventions: Drug: HS-10383
- HS-10383 Placebo (Placebo Comparator): Matching placebo to HS-10383 was administered at 8 am on the first day, 4 dose levels
  Interventions: Drug: HS-10383 Placebo

INTERVENTIONS:
Drug: HS-10383 — HS-10383 administered as one 50 mg, 150 mg, 450 mg and 900 mg tablet once daily, depending upon randomization.
  Arms: HS-10383
Drug: HS-10383 Placebo — Placebo for HS-10383
  Arms: HS-10383 Placebo

SUMMARY:
This is a first-in-human study that will investigate the safety, tolerability and pharmacokinetics of ascending single doses of HS-10383 using a randomized, double blind, placebo controlled, single center study design.

Participants in this study will receive either the study drug or placebo tablets (a placebo looks like the test drug but does not have any medicine in it). The dosage will be one single dose of study drug/placebo received on only one day. The total study duration for each participant will be usually no more than 10 days. Blood samples will be collected from the participants to monitor the safety and measure the blood level of the study drug.

DETAILED DESCRIPTION:
HS-10383 is a selective P2X3 receptor antagonist being developed for the treatment of refractory/unexplained chronic cough. This Phase 1 study will investigate the safety, tolerability and pharmacokinetics of ascending single doses of HS-10383 administered orally to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged from 18 to 45 years ;
2. Subjects need to fully understand the research content and process, as well as possible adverse reactions, and voluntarily sign the informed consent;
3. Male weight ≥ 50kg, female weight ≥ 45kg, body mass index {BMI, BMI=weight/height 2 (kg/m2)} is controlled within the range of 18~26 (including the critical value);
4. Subjects need to agree to take effective contraceptive methods from the screening date to 90 days after the last dose;
5. Male subjects must agree not to donate sperm within 90 days from the start of the administration to the last administration.

Exclusion Criteria:

1. The following medical histories, such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, metabolic endocrine system, skin disease, blood system, immune system and tumor, etc., were screened. evaluated as unsuitable to participate in this study;
2. Any known presence or history of hypogeusia, abnormal taste or dysgeusia;
3. Any known presence or history of severe allergies, or known to be allergic to the components of the test drug;
4. Use of any drugs, including prescription drugs, over-the-counter drugs or herbal preparations, cannot be avoided or expected to start 2 weeks (or 5 half-lives) before screening and throughout the study period;
5. Any findings of electrocardiogram outside from normal, such as the QT interval (QTcF) corrected by the Fridericia formula, the absolute value of QTcF for males is >450 ms, and the absolute value of QTcF for females is >470 ms;
6. Any findings of blood pressure or pulse in resting state outside from normal a: such as systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg, pulse <55 bpm or >100 bpm;
7. Serum creatinine exceeds the upper limit of normal (ULN) at screening;
8. Infectious diseases with hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody and human immunodeficiency virus (HIV) antibody test were positive at the time of screening;
9. Any findings from the medical examination (comprehensive physical examination, vital signs, blood oxygen saturation, laboratory tests, abdominal B-ultrasound and chest X-ray ) outside from normal and deemed by the investigator to be clinically significant;
10. Drug abusers, or have used soft drugs (such as marijuana) within 3 months prior to screening, or have taken hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before screening;
11. Volunteers who with a positive alcohol breath test at screening, with a history of alcohol abuse or a single consumption of more than 14 units of alcohol in the past two weeks (1 unit = 285 mL of beer, 25 mL of spirits, and 150 mL of wine);
12. Smokers or those who smoked more than 5 cigarettes per day within 3 months prior to screening, or those who could not stop using any tobacco products (including e-cigarettes) during the study;
13. Average daily intake of coffee or tea ≥ 5 cups (200mL/cup) within 3 months prior to screening;
14. Volunteers who donated or lost 250 mL more of blood in 3 months prior to screening, or had undergone major surgery in the past;
15. Volunteers who participated in any clinical trials and took any clinical trial drugs within 3 months prior to screening;
16. Difficulty swallowing solid preparations such as capsules or tablets;
17. Within 30 days prior to screening, for whatever reason, dieting or receiving dietary therapy, or major changes in dietary habits;
18. Within 30 days prior to screening and during the entire study period, consuming beverages or foods containing grapefruit (such as grapefruit, lime, star fruit, etc.), or products containing St. John's wort cannot be avoided;
19. Female subjects are pregnant or breastfeeding at the screening;
20. Females of childbearing potential with positive urine β-human chorionic gonadotropin (β-hCG) at screening, or positive serum β-hCG at baseline (day -1);
21. Volunteers who have difficulty in blood collection and cannot tolerate multiple venous blood collection and any contraindications to blood collection;
22. Volunteers who have a history of vaccination within 30 days prior to screening, or who have a vaccination plan throughout the study period;
23. As determined by the investigator, any physical or psychological disease or condition that may increase the risk of the study, affect the subject's compliance with the protocol or affect the subject's completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Evaluation | up to 9 days
  1. Adverse events (AEs), serious adverse events (SAEs) and adverse events leading to withdrawal from the study, the incidence, severity and correlation with the trial drug;
  2. Changes in laboratory tests (blood routine, urine routine, blood biochemistry and coagulation function) before and after administration;
  3. Changes in vital signs (respiration, pulse, blood pressure and body temperature) and SpO2 before and after administration;
  4. Electrocardiogram (ECG) to check the changes before and after administration.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 9 days
  To assess Cmax of single ascending oral doses of HS-10383
Time of Maximum Concentration | up to 9 days
  To assess Tmax of single ascending oral doses of HS-10383
Terminal Rate Constant | up to 9 days
  To assess λz of single ascending oral doses of HS-10383
Elimination Halflife | up to 9 days
  To assess λz of single ascending oral doses of HS-10383
Area Under the Concentration-time Curve0-t | up to 9 days
  To assess Curve0-t of single ascending oral dosCurve0-tes of HS-10383
Area Under the Concentration-time Curve0-∞ | up to 9 days
  To assess AUC0-∞ of single ascending oral doses of HS-10383
Clearance Rate | up to 9 days
  To assess Clearance Rate of single ascending oral doses of HS-10383
Apparent Volume of Distribution | up to 9 days
  To assess Vd/F of single ascending oral doses of HS-10383
Mean Retention Time | up to 9 days
  To assess MRT of single ascending oral doses of HS-10383

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Doctor, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Shandong provincial qianfoshan hospital, Jinan, Shandong, China